CLINICAL TRIAL: NCT00063661
Title: A Neuroimaging Study of Automatic Movements in Patients With Parkinson's Disease
Brief Title: Studying Automatic Movements in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030236; 03-N-0236
Record Dates: First submitted 2003-07-02; First posted 2003-07-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-05

CONDITIONS: Parkinson Disease
Keywords: fMRI; Brain Activity; Overlearned; Dual-Task; Mechanism; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease

SUMMARY:
Parkinson's disease patients usually have difficulty making automatic movements. Automatic movements are movements people often make without conscious thought.

The purpose of this study is to investigate regions of the brain that affect automatic movements and to understand the movements of Parkinson's patients. Investigators hope this knowledge will lead to better treatment for the disease.

Thirty participants will be enrolled in this study. Each will give a medical history and undergo a brief physical exam. Participants will have two MRI scans, each lasting approximately 1.5 hours. During these scans, they may be asked to move their right or left hands or to remember some letters that they have been shown. Before undergoing the second scan, participants will be asked to practice the tasks until they can perform them correctly.

DETAILED DESCRIPTION:
Patients with Parkinson's Disease (PD) are deficient in making automatic movements. The underlying neural correlates of the problem are not understood. In the present study, to investigate the brain activity contributing to this disorder, we will use specially designed dual-task paradigm and the functional magnetic resonance imaging (fMRI) technique. Thirty patients with PD will be asked to perform sequential finger-tapping movement with the right hand; results will be analyzed from 20 patients who achieve automaticity as defined in the study. In addition, we will use a dual-task paradigm to evaluate automaticity by having subjects perform either a distraction task (involving visual memory) or an interference task (tapping with the left hand) simultaneously with the sequential movements. Patients will practice to achieve automaticity. fMRI will be obtained before and after achieving automaticity. By analyzing fMRI results, we will explore the brain regions associated with deficiency of automatic movements in PD patients.

ELIGIBILITY:
INCLUSION CRITERIA:

Thirty patients with PD will be included in the study.

The diagnosis of PD is based on medical history, physical and neurological examinations, response to levodopa or dopaminergic drugs, and laboratory tests and MRI scans to exclude other diseases.

Patients will be assessed with the Unified Parkinson's Disease Rating Scale (UPDRS) and Mini-Mental State Exam (MMSE). Only patients with mild to moderate motor disability (UDRS less than or equal to 40) and without cognitive impairment (MMT score greater than or equal to 25) will be investigated.

Patients will be studied only after their medication has been withdrawn for at least 12 hours.

All subjects participating in the study should have a valid Clinical Center Medical Record Number.

The fMRI experiment will follow the standard operating procedures of the HMCS Neuroimaging Group.

EXCLUSION CRITERIA:

Subjects with psychiatric disorders or severe motor disabilities will be excluded.

Subjects with pacemakers, cardiac or neural defibrillators, intracranial aneurysm clips, intraorbital metallic structures, insulin pumps, cochlear implants, and other metallic objects will not be scanned.

Women who are pregnant are excluded from MRI because the safety of the fetus in the presence of high magnetic fields is not established. Therefore, all women of childbearing potential will have a pregnancy test performed, which must be negative, before proceeding.

Subjects under age 18 will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2003-06; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Catalan MJ, Ishii K, Honda M, Samii A, Hallett M. A PET study of sequential finger movements of varying length in patients with Parkinson's disease. Brain. 1999 Mar;122 ( Pt 3):483-95. doi: 10.1093/brain/122.3.483. PMID 10094257
- [Background] Cunnington R, Iansek R, Bradshaw JL. Movement-related potentials in Parkinson's disease: external cues and attentional strategies. Mov Disord. 1999 Jan;14(1):63-8. doi: 10.1002/1531-8257(199901)14:13.0.co;2-v. PMID 9918346
- [Background] Catalan MJ, Honda M, Weeks RA, Cohen LG, Hallett M. The functional neuroanatomy of simple and complex sequential finger movements: a PET study. Brain. 1998 Feb;121 ( Pt 2):253-64. doi: 10.1093/brain/121.2.253. PMID 9549504